CLINICAL TRIAL: NCT03850314
Title: The Effects of Glycine on Atherosclerosis and Metabolic Syndrome-related Parameters: A Clinical and Ex-vivo Study.
Brief Title: The Effects of Glycine on Atherosclerosis and Metabolic Syndrome-related Parameters.
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Prof. Tony hayek MD (Other)
Responsible Party: Sponsor-Investigator, Prof. Tony hayek MD, Director, Department of Internal Medicine "E"., Rambam Health Care Campus
Organization: Rambam Health Care Campus (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RMB-18-0621
Record Dates: First submitted 2019-02-19; First posted 2019-02-21 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Metabolic Syndrome; Dyslipidemias; Diabetes Mellitus; Obesity; Atherosclerosis
MeSH Terms: conditions — Metabolic Syndrome; Dyslipidemias; Diabetes Mellitus; Obesity; Atherosclerosis | interventions — Glycine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Glycine (Experimental): Glycine total daily dose of 150mg/kg divided three times daily with meals (powder dissolved in 1 cup of water) for 12 weeks.
  Interventions: Dietary Supplement: Glycine

INTERVENTIONS:
Dietary Supplement: Glycine — Glycine powder to be dissolved in water.

SUMMARY:
The current study will test the central hypothesis that Glycine supplementation in humans improves Lipid profile and therefore reduces the risk of Atherosclerosis. Secondary outcomes including Insulin sensitivity and parameters related to Metabolic Syndrome (MetS) will also be measured. Furthermore, a mechanistic study in an ex-vivo model will test the hypothesis that Glycine via its key biosynthetic pathway involving Serine Hydroxymethyltransferase 2 (SHMT2), is athero-protective by inhibiting Sterol regulatory element-binding protein 2 (SREBP2)-mediated cholesterol biosynthesis in murine macrophage-like cell line.

ELIGIBILITY:
Inclusion Criteria:

* Male between the ages of 40-65 years old.
* Fulfill at least three of the five diagnostic criteria for the Metabolic Syndrome.
* To be able to give their written consent to participate in this study.

Exclusion Criteria:

* Abnormal Liver function tests ≥ 3 times upper limit of normal (ULN).
* Chronic liver disease other than NAFLD.
* Previous gastric or small bowel surgery.
* Abnormal Thyroid-stimulating hormone (TSH) level.
* Known Tobacco Smoking more than 10 cigarettes per day.
* Known alcohol consumption more than 2 drink per day.
* Use of medications that include: Insulin or Insulin secretagogues, Thiazolidinediones, Glucocorticosteroids, Hormone replacement therapy.
* Fever > 38.2 °C in the past 2 weeks.
* Autoimmune or Auto-inflammatory disease.
* Chronic kidney disease ≥ stage III.
* Nephrotic syndrome.
* Hemoglobin <12 g/dL.
* Metal clips or implants that preclude magnetic resonance imaging.

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-03 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
LDL Cholesterol levels | 12 weeks
  Change in LDL Cholesterol levels

SECONDARY OUTCOMES:
Triglyceride levels | 12 weeks
  Change in Triglyceride levels
HDL Cholesterol levels | 12 weeks
  Change in HDL Cholesterol levels
HbA1C levels | 12 weeks
  Change in Glycated hemoglobin (HbA1C) levels

CONTACTS AND LOCATIONS:
Overall Officials: Tony Hayek, MD, Principal Investigator — Rambam Health Care Campus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moore KJ, Sheedy FJ, Fisher EA. Macrophages in atherosclerosis: a dynamic balance. Nat Rev Immunol. 2013 Oct;13(10):709-21. doi: 10.1038/nri3520. Epub 2013 Sep 2. PMID 23995626
- [Background] Weber C, Noels H. Atherosclerosis: current pathogenesis and therapeutic options. Nat Med. 2011 Nov 7;17(11):1410-22. doi: 10.1038/nm.2538. PMID 22064431
- [Background] Michas G, Micha R, Zampelas A. Dietary fats and cardiovascular disease: putting together the pieces of a complicated puzzle. Atherosclerosis. 2014 Jun;234(2):320-8. doi: 10.1016/j.atherosclerosis.2014.03.013. Epub 2014 Mar 27. PMID 24727233
- [Background] Sacks FM, Lichtenstein AH, Wu JHY, Appel LJ, Creager MA, Kris-Etherton PM, Miller M, Rimm EB, Rudel LL, Robinson JG, Stone NJ, Van Horn LV; American Heart Association. Dietary Fats and Cardiovascular Disease: A Presidential Advisory From the American Heart Association. Circulation. 2017 Jul 18;136(3):e1-e23. doi: 10.1161/CIR.0000000000000510. Epub 2017 Jun 15. PMID 28620111
- [Background] Rom O, Aviram M. It is not just lipids: proatherogenic vs. antiatherogenic roles for amino acids in macrophage foam cell formation. Curr Opin Lipidol. 2017 Feb;28(1):85-87. doi: 10.1097/MOL.0000000000000377. No abstract available. PMID 28030455
- [Background] Shah SH, Bain JR, Muehlbauer MJ, Stevens RD, Crosslin DR, Haynes C, Dungan J, Newby LK, Hauser ER, Ginsburg GS, Newgard CB, Kraus WE. Association of a peripheral blood metabolic profile with coronary artery disease and risk of subsequent cardiovascular events. Circ Cardiovasc Genet. 2010 Apr;3(2):207-14. doi: 10.1161/CIRCGENETICS.109.852814. Epub 2010 Feb 19. PMID 20173117
- [Background] Wurtz P, Raiko JR, Magnussen CG, Soininen P, Kangas AJ, Tynkkynen T, Thomson R, Laatikainen R, Savolainen MJ, Laurikka J, Kuukasjarvi P, Tarkka M, Karhunen PJ, Jula A, Viikari JS, Kahonen M, Lehtimaki T, Juonala M, Ala-Korpela M, Raitakari OT. High-throughput quantification of circulating metabolites improves prediction of subclinical atherosclerosis. Eur Heart J. 2012 Sep;33(18):2307-16. doi: 10.1093/eurheartj/ehs020. Epub 2012 Mar 26. PMID 22450427
- [Background] Bhattacharya S, Granger CB, Craig D, Haynes C, Bain J, Stevens RD, Hauser ER, Newgard CB, Kraus WE, Newby LK, Shah SH. Validation of the association between a branched chain amino acid metabolite profile and extremes of coronary artery disease in patients referred for cardiac catheterization. Atherosclerosis. 2014 Jan;232(1):191-6. doi: 10.1016/j.atherosclerosis.2013.10.036. Epub 2013 Nov 12. PMID 24401236
- [Background] Yang R, Dong J, Zhao H, Li H, Guo H, Wang S, Zhang C, Wang S, Wang M, Yu S, Chen W. Association of branched-chain amino acids with carotid intima-media thickness and coronary artery disease risk factors. PLoS One. 2014 Jun 9;9(6):e99598. doi: 10.1371/journal.pone.0099598. eCollection 2014. PMID 24910999
- [Background] Yang RY, Wang SM, Sun L, Liu JM, Li HX, Sui XF, Wang M, Xiu HL, Wang S, He Q, Dong J, Chen WX. Association of branched-chain amino acids with coronary artery disease: A matched-pair case-control study. Nutr Metab Cardiovasc Dis. 2015 Oct;25(10):937-42. doi: 10.1016/j.numecd.2015.06.003. Epub 2015 Jun 14. PMID 26231617
- [Background] Grajeda-Iglesias C, Aviram M. Specific Amino Acids Affect Cardiovascular Diseases and Atherogenesis via Protection against Macrophage Foam Cell Formation: Review Article. Rambam Maimonides Med J. 2018 Jul 30;9(3):e0022. doi: 10.5041/RMMJ.10337. PMID 29944113
- [Background] Ding Y, Svingen GF, Pedersen ER, Gregory JF, Ueland PM, Tell GS, Nygard OK. Plasma Glycine and Risk of Acute Myocardial Infarction in Patients With Suspected Stable Angina Pectoris. J Am Heart Assoc. 2015 Dec 31;5(1):e002621. doi: 10.1161/JAHA.115.002621. PMID 26722126
- [Background] Rom O, Aviram M. Endogenous or exogenous antioxidants vs. pro-oxidants in macrophage atherogenicity. Curr Opin Lipidol. 2016 Apr;27(2):204-6. doi: 10.1097/MOL.0000000000000287. No abstract available. PMID 26959710
- [Background] Rom O, Grajeda-Iglesias C, Najjar M, Abu-Saleh N, Volkova N, Dar DE, Hayek T, Aviram M. Atherogenicity of amino acids in the lipid-laden macrophage model system in vitro and in atherosclerotic mice: a key role for triglyceride metabolism. J Nutr Biochem. 2017 Jul;45:24-38. doi: 10.1016/j.jnutbio.2017.02.023. Epub 2017 Apr 6. PMID 28431321
- [Background] Yan-Do R, MacDonald PE. Impaired "Glycine"-mia in Type 2 Diabetes and Potential Mechanisms Contributing to Glucose Homeostasis. Endocrinology. 2017 May 1;158(5):1064-1073. doi: 10.1210/en.2017-00148. PMID 28323968
- [Background] Yamakado M, Tanaka T, Nagao K, Ishizaka Y, Mitushima T, Tani M, Toda A, Toda E, Okada M, Miyano H, Yamamoto H. Plasma amino acid profile is associated with visceral fat accumulation in obese Japanese subjects. Clin Obes. 2012 Feb;2(1-2):29-40. doi: 10.1111/j.1758-8111.2012.00039.x. Epub 2012 May 22. PMID 25586045
- [Background] Gaggini M, Carli F, Rosso C, Buzzigoli E, Marietti M, Della Latta V, Ciociaro D, Abate ML, Gambino R, Cassader M, Bugianesi E, Gastaldelli A. Altered amino acid concentrations in NAFLD: Impact of obesity and insulin resistance. Hepatology. 2018 Jan;67(1):145-158. doi: 10.1002/hep.29465. Epub 2017 Nov 17. PMID 28802074
- [Background] Mirmiran P, Bahadoran Z, Ghasemi A, Azizi F. Contribution of dietary amino acids composition to incidence of cardiovascular outcomes: A prospective population-based study. Nutr Metab Cardiovasc Dis. 2017 Jul;27(7):633-641. doi: 10.1016/j.numecd.2017.05.003. Epub 2017 May 15. PMID 28684082
- [Background] Petrat F, Boengler K, Schulz R, de Groot H. Glycine, a simple physiological compound protecting by yet puzzling mechanism(s) against ischaemia-reperfusion injury: current knowledge. Br J Pharmacol. 2012 Apr;165(7):2059-72. doi: 10.1111/j.1476-5381.2011.01711.x. PMID 22044190
- [Background] Razak MA, Begum PS, Viswanath B, Rajagopal S. Multifarious Beneficial Effect of Nonessential Amino Acid, Glycine: A Review. Oxid Med Cell Longev. 2017;2017:1716701. doi: 10.1155/2017/1716701. Epub 2017 Mar 1. PMID 28337245
- [Background] McCarty MF, Barroso-Aranda J, Contreras F. The hyperpolarizing impact of glycine on endothelial cells may be anti-atherogenic. Med Hypotheses. 2009 Aug;73(2):263-4. doi: 10.1016/j.mehy.2008.12.021. Epub 2009 Feb 18. PMID 19232835
- [Background] McCarty MF, DiNicolantonio JJ. The cardiometabolic benefits of glycine: Is glycine an 'antidote' to dietary fructose? Open Heart. 2014 May 28;1(1):e000103. doi: 10.1136/openhrt-2014-000103. eCollection 2014. No abstract available. PMID 25332814
- [Background] Wang W, Wu Z, Dai Z, Yang Y, Wang J, Wu G. Glycine metabolism in animals and humans: implications for nutrition and health. Amino Acids. 2013 Sep;45(3):463-77. doi: 10.1007/s00726-013-1493-1. Epub 2013 Apr 25. PMID 23615880
- [Background] Morscher RJ, Ducker GS, Li SH, Mayer JA, Gitai Z, Sperl W, Rabinowitz JD. Mitochondrial translation requires folate-dependent tRNA methylation. Nature. 2018 Feb 1;554(7690):128-132. doi: 10.1038/nature25460. Epub 2018 Jan 24. PMID 29364879
- [Background] Mardinoglu A, Agren R, Kampf C, Asplund A, Uhlen M, Nielsen J. Genome-scale metabolic modelling of hepatocytes reveals serine deficiency in patients with non-alcoholic fatty liver disease. Nat Commun. 2014;5:3083. doi: 10.1038/ncomms4083. PMID 24419221
- [Background] Kruth HS. Macrophage foam cells and atherosclerosis. Front Biosci. 2001 Mar 1;6:D429-55. doi: 10.2741/kruth. PMID 11229875
- [Background] Diaz-Flores M, Cruz M, Duran-Reyes G, Munguia-Miranda C, Loza-Rodriguez H, Pulido-Casas E, Torres-Ramirez N, Gaja-Rodriguez O, Kumate J, Baiza-Gutman LA, Hernandez-Saavedra D. Oral supplementation with glycine reduces oxidative stress in patients with metabolic syndrome, improving their systolic blood pressure. Can J Physiol Pharmacol. 2013 Oct;91(10):855-60. doi: 10.1139/cjpp-2012-0341. Epub 2013 Jun 17. PMID 24144057
- [Background] Heresco-Levy U, Javitt DC, Ermilov M, Mordel C, Silipo G, Lichtenstein M. Efficacy of high-dose glycine in the treatment of enduring negative symptoms of schizophrenia. Arch Gen Psychiatry. 1999 Jan;56(1):29-36. doi: 10.1001/archpsyc.56.1.29. PMID 9892253
- [Background] Evins AE, Fitzgerald SM, Wine L, Rosselli R, Goff DC. Placebo-controlled trial of glycine added to clozapine in schizophrenia. Am J Psychiatry. 2000 May;157(5):826-8. doi: 10.1176/appi.ajp.157.5.826. PMID 10784481
- [Background] Mardinoglu A, Bjornson E, Zhang C, Klevstig M, Soderlund S, Stahlman M, Adiels M, Hakkarainen A, Lundbom N, Kilicarslan M, Hallstrom BM, Lundbom J, Verges B, Barrett PH, Watts GF, Serlie MJ, Nielsen J, Uhlen M, Smith U, Marschall HU, Taskinen MR, Boren J. Personal model-assisted identification of NAD+ and glutathione metabolism as intervention target in NAFLD. Mol Syst Biol. 2017 Mar 2;13(3):916. doi: 10.15252/msb.20167422. PMID 28254760
- [Background] National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults (Adult Treatment Panel III). Third Report of the National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults (Adult Treatment Panel III) final report. Circulation. 2002 Dec 17;106(25):3143-421. No abstract available. PMID 12485966
- [Background] Wallace TM, Levy JC, Matthews DR. Use and abuse of HOMA modeling. Diabetes Care. 2004 Jun;27(6):1487-95. doi: 10.2337/diacare.27.6.1487. PMID 15161807
- [Background] Dulai PS, Sirlin CB, Loomba R. MRI and MRE for non-invasive quantitative assessment of hepatic steatosis and fibrosis in NAFLD and NASH: Clinical trials to clinical practice. J Hepatol. 2016 Nov;65(5):1006-1016. doi: 10.1016/j.jhep.2016.06.005. Epub 2016 Jun 14. PMID 27312947
- [Background] Permutt Z, Le TA, Peterson MR, Seki E, Brenner DA, Sirlin C, Loomba R. Correlation between liver histology and novel magnetic resonance imaging in adult patients with non-alcoholic fatty liver disease - MRI accurately quantifies hepatic steatosis in NAFLD. Aliment Pharmacol Ther. 2012 Jul;36(1):22-9. doi: 10.1111/j.1365-2036.2012.05121.x. Epub 2012 May 3. PMID 22554256